CLINICAL TRIAL: NCT00907946
Title: A Prospective, Randomized Trial Comparing Previously Placed Nephrostomy Tract and Single Stage Percutaneous Nephrolithotomy and Its Effects on Infection and Bleeding Related Complications
Brief Title: Comparing Previously Placed Nephrostomy Tract (NT) Versus Single Stage Percutaneous Nephrolithotomy (PCNL)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Alana Desai PCNL Study-09-0709
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Urolithiasis
Keywords: Renal stones
MeSH Terms: conditions — Urolithiasis; Nephrolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NT prior to PCNL (Experimental): A bladder urine culture will be obtained prior to nephrostomy tube placement and antibiotic treatment will be initiated if necessary. A nephrostomy tube will be placed at least one week prior to surgery in the Vascular Interventional Radiology (VIR) suite under fluoroscopic or ultrasound guidance. The type of imaging will be determined by the radiologist at the time of procedure and documented. A renal pelvis urine culture will be obtained at the time of nephrostomy tube placement. If the culture is positive, the patients will be treated with appropriate antibiotics for at least one week prior to PCNL. If the culture is negative, the patient will be stratified into 2 groups:
  1. Hydronephrosis present and/or stone greater than 2cm empiric antibiotics will be initiated.
  2. If neither of the above criteria (a.) are met, and the urine culture is negative, no antibiotics will be administered except peri-operatively according to standard protocol.
  Interventions: Procedure: NT 1 day before PCNL
- NT at the surgery (No Intervention): A bladder urine culture will be obtained prior to surgery and appropriate antibiotic treatment will be initiated if necessary. The nephrostomy tract will be placed at the time of surgery under fluoroscopic guidance. All patients will receive empiric intravenous peri-operative antibiotics at induction. Renal pelvis urine and stone will be collected for culture and post-operative treatment will be initiated if necessary.

INTERVENTIONS:
Procedure: NT 1 day before PCNL — A bladder urine culture will be obtained prior to nephrostomy tube placement and antibiotic treatment will be initiated if necessary. A nephrostomy tube will be placed at least one day prior to surgery in the Vascular Interventional Radiology (VIR) suite under fluoroscopic or ultrasound guidance. The type of imaging will be determined by the radiologist at the time of procedure and documented. A renal pelvis urine culture will be obtained at the time of nephrostomy tube placement. If the culture is positive, the patients will be treated with appropriate antibiotics for at least one week prior to PCNL. If the culture is negative, the patient will be stratified into 2 groups:
  1. Hydronephrosis present and/or stone greater than 2cm empiric antibiotics will be initiated.
  2. If neither of the above criteria (a.) are met, and the urine culture is negative, no antibiotics will be administered except peri-operatively according to standard protocol.
  Arms: NT prior to PCNL

SUMMARY:
The investigators are trying to determine whether placement of a nephrostomy tube prior to definitive stone surgery and under ultrasonic or fluoroscopic guidance will reduce complications related to bleeding and infection compare to obtaining renal access at the time of surgery.

DETAILED DESCRIPTION:
We seek to identify whether the placement of a nephrostomy tract prior to surgery versus at the time of PCNL will: 1. decrease blood loss and related complications, and 2. decrease infection-related complications by providing the ability to an accurate collection of urine for culture and initiating appropriate antibiotic treatment prior to definitive stone management. In addition, we seek to determine whether renal puncture under fluoroscopic vs ultrasonic guidance is associated with less blood loss. Although retrospective studies have shown some benefit to placing the nephrostomy tube prior to surgery in terms of decreased blood loss, there are no well-designed, prospective studies comparing the two treatment approaches. We seek to determine which treatment approach is safer, more efficacious, and more cost-effective through a prospective, randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years to 90 years old,
* Patients with stone disease
* Patients who hoose to have PCNL for treatment
* Patients who understand the informed consent

Exclusion Criteria:

* Minors
* Unable to understand the informed consent
* Unwilling to fill out the SF 36 questionnaire

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Reduction of complications related to bleeding and infection | 3 years
  We aim to determine whether placement of a nephrostomy tube prior to definitive stone surgery and under ultrasonic or fluoroscopic guidance will reduce complications related to bleeding and infection compared to obtaining renal access at the time of surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States